CLINICAL TRIAL: NCT01434537
Title: Venepuncture and Vein Cannulation With Support of the AccuVein AV300 Vein Scanner in Paediatric Patients in a Pre-operation Setting
Brief Title: Evaluation of a Touchless Vein Scanner for Venepuncture and Cannulation in Pediatric Patients
Acronym: VENSCAN
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Prof. , MD Director of the Department of Anaesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany
Other Study IDs: VENSCAN
Record Dates: First submitted 2011-07-29; First posted 2011-09-15 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Venepuncture
Keywords: pediatric anesthesia; venepuncture; peripheral venous access

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SCAN: Venepuncture performed with support of the AccuVein 300 vein scanner.
- NO_SCAN: Venepuncture without support of the vein scanner.

SUMMARY:
Evaluation of the AccuVein ® AV 300 vein scanner in clinical routine in a pediatric operation room setting for a 4 weeks period. Assessment of usability, anonymous clinical register of every venepuncture(age, gender, size, weight, punction site, number of attempts, time until successful cannulation, local anaesthesia, general anaesthesia, pain scales: faces pain scale und BPS/BPOS).

DETAILED DESCRIPTION:
For application of drugs and liquids a peripheral venous access is necessary in anaesthesiological procedures.The peripheral venepuncture is a painful procedure and induces a higher level of perioperative stress in children.

The punction of peripheral veins in children can be made difficult by the often distinctive amount of subcutaneous fat or other medical conditions.

The AccuVein ® AV300 vein scanner is a contactless, laser-driven device made for facilitate the search for peripheral veins up to a depth of 7mm. This could lead to a minimization of time until successful puncture and smaller number of failures.

ELIGIBILITY:
Inclusion Criteria:

* age from 0 to 17 years
* perioperative indication for peripheral venous access
* regular work time of the operation room from 7 am to 4 pm

Exclusion Criteria:

* age more than 17 years
* no indication for or already established venous access

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients from 0 to 17 years in a peripoerative setting in the pediatric operation room with need for peripheral venous access.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
time until completion of procedure | Day 1
  minutes until successful puncture and cannulation of peripheral vein

SECONDARY OUTCOMES:
number of attempts until completion of procedure | Day 1
  number of attempts until successful puncture and cannulation of peripheral vein

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum and Campus Charité Mitte, Charité - Universitaetsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Rothbart A, Yu P, Muller-Lobeck L, Spies CD, Wernecke KD, Nachtigall I. Peripheral intravenous cannulation with support of infrared laser vein viewing system in a pre-operation setting in pediatric patients. BMC Res Notes. 2015 Sep 21;8:463. doi: 10.1186/s13104-015-1431-2. PMID 26391665